CLINICAL TRIAL: NCT01134562
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Assess the Safety and Tolerability of Single Ascending Doses of KAI-4169 in Hemodialysis Subjects With Secondary Hyperparathyroidism
Brief Title: Safety, Tolerability and Pharmacokinetics of Etelcalcetide in Hemodialysis Patients With Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KAI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: KAI-4169-002; 20130139 (Other: Amgen, Inc)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-05

CONDITIONS: Hyperparathyroidism, Secondary
Keywords: Clinical Trial, Phase 1; Renal Dialysis; Secondary Hyperparathyroidism; Parathyroid hormone
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received a single dose of placebo intravenous (IV) injection after hemodialysis.
  Interventions: Drug: Placebo
- Etelcalcetide (Experimental): Participants received a single dose of etelcalcetide by intravenous (IV) injection after hemodialysis.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Placebo — Single IV injection.
  Arms: Placebo
Drug: Etelcalcetide — Single IV injection. The initial dose was 5 mg and dose escalation proceeded with subsequent doses of 10 mg, 20 mg, 40 mg and 60 mg.
  Other Names: KAI-4169; AMG 416
  Arms: Etelcalcetide

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of single rising doses of etelcalcetide in hemodialysis patients with secondary hyperparathyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Subjects provides written informed consent.
* Intact parathyroid hormone (iPTH) ≥ 400 pg/mL (≥ 300 and < 1200 pg/ml for Cohorts 1-3).
* Serum corrected calcium ≥ 9.0 mg/dL
* Receiving hemodialysis three times per week for at least 3 months and had adequate hemodialysis with a delivered Kt/V (dialyzer clearance of urea * dialysis time/ volume of distribution of urea) ≥ 1.2 or urea reduction ratio (URR)

  ≥ 65%.
* Excepting chronic renal failure, subject is judged to be in stable medical condition based on medical history, physical examination, and routine laboratory tests

Exclusion Criteria:

* History or symptomatic ventricular dysrhythmias
* History of angina pectoris or congestive heart failure
* History of myocardial infarction, coronary angioplasty, or coronary artery bypass grafting within the past 6 months
* History of or treatment for seizure disorder
* Recent (3 months) parathyroidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09-07; Primary Completion 2011-04-02 (Actual); Study Completion 2011-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Bell, MD, Study Director — KAI Pharmaceuticals
Locations (5):
- United States (3):
  - Cypress, California
  - Shreveport, Louisiana
  - Houston, Texas
- Australia (2):
  - Brisbane, Queensland
  - Melbourne, Victoria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 1 center in Australia and 2 centers in the United States from 07 September 2010 to 02 April 2011.
Pre-assignment Details: Cohorts 1-3 were conducted with a two-period crossover design. Each cohort enrolled four participants randomized 1:1 to etelcalcetide followed by placebo or placebo followed by etelcalcetide. Cohorts 4 and 5 followed a parallel group design. Within each cohort eight participants were randomized 1:1 to receive placebo or etelcalcetide.
Groups:
- Cohort 1: Placebo/Etelcalcetide 5 mg: Participants in Cohort 1 received single doses of 5 mg etelcalcetide and placebo in a crossover design, 7-14 days apart
- Cohort 2: Placebo/Etelcalcetide 10 mg: Participants in Cohort 2 received single doses of 10 mg etelcalcetide and placebo in a crossover design, 7-14 days apart
- Cohort 3: Placebo/Etelcalcetide 20 mg: Participants in Cohort 3 received single doses of 20 mg etelcalcetide and placebo in a crossover design, 7-14 days apart
- Cohort 4: Placebo/Etelcalcetide 40 mg: Participants in Cohort 4 received a single dose of 40 mg etelcalcetide or placebo in a parallel group design.
- Cohort 5: Placebo/Etelcalcetide 60 mg: Participants in Cohort 5 received a single dose of 60 mg etelcalcetide or placebo in a parallel group design.
Period: Overall Study
Arm/Group | Cohort 1: Placebo/Etelcalcetide 5 mg | Cohort 2: Placebo/Etelcalcetide 10 mg | Cohort 3: Placebo/Etelcalcetide 20 mg | Cohort 4: Placebo/Etelcalcetide 40 mg | Cohort 5: Placebo/Etelcalcetide 60 mg
Started | 4 | 4 | 4 | 8 | 8
Completed | 4 | 3 | 4 | 8 | 8
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Placebo/Etelcalcetide 5 mg | Cohort 2: Placebo/Etelcalcetide 10 mg | Cohort 3: Placebo/Etelcalcetide 20 mg | Cohort 4: Placebo/Etelcalcetide 40 mg | Cohort 5: Placebo/Etelcalcetide 60 mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 8 | 8 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (10.4) | 59.0 (14.5) | 52.8 (21.2) | 52.9 (14.6) | 47.5 (10.9) | 52.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 4 | 2 | 8
  Male | 3 | 4 | 3 | 4 | 6 | 20
Race [Count of Participants; unit: Participants]
  White | 1 | 0 | 1 | 0 | 1 | 3
  African American | 2 | 4 | 3 | 8 | 7 | 24
  Asian | 1 | 0 | 0 | 0 | 0 | 1
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Non-Hispanic or Latino | 4 | 4 | 4 | 8 | 8 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: For Cohorts 1 to 3, from administration of study drug up until 21 days after study drug administration; for Cohorts 4 and 5 from administration of study drug until 28 days after study drug administration.
Population: All participants who were randomized and received any amount of study medication.
Measure: Number; unit: participants
Groups:
- Pooled Placebo: Participants received a single dose of placebo intravenous (IV) injection after hemodialysis.
- Etelcalcetide 5 mg: Participants received a single dose of 5 mg etelcalcetide IV injection after hemodialysis.
- Etelcalcetide 10 mg: Participants received a single dose of 10 mg etelcalcetide IV injection after hemodialysis.
- Etelcalcetide 20 mg: Participants received a single dose of 20 mg etelcalcetide IV injection after hemodialysis.
- Etelcalcetide 40 mg: Participants received a single dose of 40 mg etelcalcetide IV injection after hemodialysis.
- Etelcalcetide 60 mg: Participants received a single dose of 60 mg etelcalcetide IV injection after hemodialysis.
Arm/Group | Pooled Placebo | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide 20 mg | Etelcalcetide 40 mg | Etelcalcetide 60 mg
Number analyzed (Participants) | 20 | 4 | 3 | 4 | 4 | 4
participants
  Any adverse events | 2 | 1 | 1 | 1 | 4 | 2
  Serious adverse events | 1 | 0 | 0 | 0 | 0 | 0
  Withdrawal due to adverse events | 1 | 0 | 0 | 0 | 0 | 0
  Deaths due to adverse events | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related adverse events | 1 | 1 | 1 | 0 | 4 | 2

2. Secondary Outcome: Percent Change From Baseline in Serum Parathyroid Hormone (PTH)
Time Frame: Baseline and 30 minutes, 1, 4, 8, 18, 24, 32, 42, 48, and 56 hours post-dose, day 4 (discharge) and for Cohorts 4 and 5 only, days 8, 15 and 29
Population: Participants who were randomized and received any amount of study medication with available data at each time point. Only participants in Cohorts 4 and 5 had PTH assessed on days 8, 15 and 29.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Pooled Placebo: Participants received a single dose of placebo IV injection after hemodialysis.
Arm/Group | Pooled Placebo | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide 20 mg | Etelcalcetide 40 mg | Etelcalcetide 60 mg
Number analyzed (Participants) | 20 | 4 | 3 | 4 | 4 | 4
percent change
  30 Minutes | 1.381 (20.429) | -63.179 (5.135) | -68.890 (9.616) | -70.021 (11.273) | -72.435 (11.176) | -77.471 (5.979)
  1 Hour | -0.540 (17.092) | -64.094 (4.547) | -73.060 (7.959) | -70.309 (9.601) | -75.898 (11.333) | -78.757 (4.921)
  4 Hours | 3.922 (30.491) | -39.975 (14.961) | -51.734 (23.294) | -72.893 (14.821) | -74.627 (13.479) | -80.266 (7.476)
  8 Hours | 4.014 (25.061) | -39.789 (9.694) | -52.075 (16.841) | -70.904 (15.663) | -77.031 (8.236) | -84.184 (6.461)
  18 Hours | -13.552 (25.000) | -23.751 (10.615) | -48.744 (15.460) | -72.653 (16.154) | -78.332 (7.393) | -85.547 (6.056)
  24 Hours | -16.888 (30.497) | -23.420 (10.289) | -46.642 (18.136) | -41.723 (26.353) | -77.206 (4.005) | -84.845 (6.208)
  32 Hours | -16.434 (34.774) | -18.406 (15.484) | -32.987 (26.492) | -55.919 (33.153) | -69.795 (4.812) | -83.439 (5.802)
  42 Hours | -20.394 (25.119) | -9.087 (10.439) | -34.912 (22.835) | -57.207 (32.894) | -63.258 (5.239) | -76.096 (9.079)
  48 Hours | -21.664 (28.956) | -14.905 (16.588) | -36.142 (24.957) | -43.145 (43.175) | -55.486 (1.761) | -71.268 (11.557)
  56 Hours: number analyzed (Participants) | 20 | 3 | 3 | 4 | 4 | 4
  56 Hours | -15.484 (33.626) | -2.968 (20.870) | -21.994 (34.015) | -43.271 (44.442) | -48.128 (3.740) | -60.112 (16.074)
  Day 4-Discharge | -11.192 (33.131) | -7.428 (15.016) | 13.264 (23.682) | -48.533 (32.739) | -49.277 (6.274) | -62.628 (12.335)
  Day 8: number analyzed (Participants) | 8 | 0 | 0 | 0 | 4 | 4
  Day 8 | -31.881 (38.536) |  |  |  | -30.766 (32.248) | -61.093 (5.804)
  Day 15: number analyzed (Participants) | 8 | 0 | 0 | 0 | 4 | 4
  Day 15 | -33.993 (44.928) |  |  |  | -34.149 (22.536) | -58.510 (15.169)
  Day 29: number analyzed (Participants) | 8 | 0 | 0 | 0 | 4 | 4
  Day 29 | -31.394 (47.249) |  |  |  | -14.750 (28.303) | -44.478 (16.631)

3. Secondary Outcome: Percent Change From Baseline in Serum Corrected Calcium
Time Frame: as for outcome 2
Population: Participants who were randomized and received any amount of study medication and with available data at each time point. Only participants in Cohorts 4 and 5 had serum corrected calcium assessed on days 8, 15 and 29.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pooled Placebo | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide 20 mg | Etelcalcetide 40 mg | Etelcalcetide 60 mg
Number analyzed (Participants) | 20 | 4 | 3 | 4 | 4 | 4
percent change
  30 Minutes: number analyzed (Participants) | 19 | 4 | 3 | 4 | 4 | 4
  30 Minutes | 0.024 (3.881) | 0.106 (4.550) | -2.883 (2.457) | -2.589 (1.665) | -0.572 (2.126) | 1.951 (6.723)
  1 Hour | -0.295 (4.644) | 0.256 (1.043) | -5.176 (2.874) | -2.574 (1.335) | -3.700 (3.395) | 3.445 (9.876)
  4 Hours | 0.540 (4.998) | -3.427 (1.201) | -7.795 (2.473) | -5.515 (1.939) | -3.599 (2.991) | -1.258 (10.241)
  8 Hours | 0.945 (5.894) | -5.533 (8.724) | -10.697 (4.257) | -7.685 (2.633) | -5.895 (5.393) | -4.057 (10.732)
  18 Hours | 3.669 (7.885) | -3.103 (3.399) | -8.018 (6.150) | -9.560 (4.703) | -5.993 (9.270) | -5.738 (10.402)
  24 Hours | 3.853 (8.667) | -3.003 (4.149) | -8.826 (2.766) | -11.436 (5.463) | -8.436 (10.582) | -5.688 (9.762)
  32 Hours | 3.079 (9.187) | -1.632 (7.315) | -9.436 (2.192) | -10.644 (8.525) | -6.155 (12.748) | -7.146 (10.382)
  42 Hours | 3.209 (9.716) | -4.815 (8.629) | -9.049 (3.745) | -11.700 (8.151) | -9.186 (8.793) | -9.082 (7.392)
  48 Hours | 2.918 (8.965) | -2.781 (7.855) | -9.115 (0.280) | -9.458 (7.873) | -8.174 (9.005) | -10.911 (9.479)
  56 Hours: number analyzed (Participants) | 20 | 3 | 3 | 4 | 4 | 4
  56 Hours | 1.920 (10.339) | -1.583 (4.258) | -10.338 (4.119) | -9.227 (6.946) | -8.970 (8.789) | -12.300 (9.491)
  Day 4-Discharge | 1.556 (10.240) | -2.577 (12.131) | -7.405 (4.208) | -9.200 (6.760) | -8.180 (9.334) | -13.186 (9.781)
  Day 8: number analyzed (Participants) | 8 | 0 | 0 | 0 | 4 | 4
  Day 8 | 0.632 (10.506) |  |  |  | -3.985 (12.631) | -8.859 (3.740)
  Day 15: number analyzed (Participants) | 8 | 0 | 0 | 0 | 4 | 4
  Day 15 | 3.827 (8.196) |  |  |  | -0.238 (8.371) | -6.885 (9.669)
  Day 29: number analyzed (Participants) | 8 | 0 | 0 | 0 | 4 | 4
  Day 29 | 4.228 (9.346) |  |  |  | 2.221 (2.378) | 3.620 (7.196)

4. Secondary Outcome: Percent Change From Baseline in Ionized Calcium
Time Frame: Baseline and 30 minutes, 1, 4, 8, 18, 24, 32, 42, 48, and 56 hours post-dose, and day 4 (discharge).
Population: Participants who were randomized and received any amount of study medication with available data at each time point
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pooled Placebo | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide 20 mg | Etelcalcetide 40 mg | Etelcalcetide 60 mg
Number analyzed (Participants) | 20 | 4 | 3 | 4 | 4 | 3
percent change
  30 Minutes | -0.118 (2.920) | 0.234 (2.172) | -2.940 (4.619) | -0.122 (2.400) | -0.934 (2.007) | -3.300 (5.716)
  1 Hour: number analyzed (Participants) | 20 | 4 | 3 | 4 | 3 | 3
  1 Hour | -0.151 (2.577) | -1.406 (3.173) | -1.394 (3.841) | -0.442 (4.233) | -3.072 (7.850) | 1.595 (1.118)
  4 Hours | 0.744 (3.126) | -3.436 (4.124) | -6.015 (1.847) | -3.550 (4.054) | -3.759 (11.275) | -1.514 (3.049)
  8 Hours | 1.924 (4.128) | -0.703 (4.896) | -6.218 (2.395) | -7.160 (6.947) | -3.867 (10.572) | -8.652 (3.231)
  18 Hours | 6.570 (5.729) | -2.168 (4.508) | -4.125 (3.667) | -6.571 (5.425) | -3.949 (5.644) | -12.139 (5.122)
  24 Hours | 6.920 (6.835) | -0.663 (3.640) | -3.822 (3.953) | -7.093 (8.308) | -5.395 (11.404) | -10.916 (4.793)
  32 Hours | 5.925 (7.251) | 0.918 (3.431) | -2.830 (5.873) | -4.044 (11.718) | -5.090 (10.317) | -7.627 (2.563)
  42 Hours | 8.157 (8.080) | -0.456 (3.392) | -4.213 (1.195) | -5.980 (8.479) | -3.212 (6.593) | -12.00 (3.337)
  48 Hours | 6.080 (8.323) | -1.376 (4.136) | -2.919 (3.392) | -5.282 (9.031) | -2.468 (9.489) | -13.449 (3.961)
  56 Hours: number analyzed (Participants) | 20 | 3 | 3 | 4 | 4 | 3
  56 Hours | 5.991 (7.704) | 0.612 (5.530) | -3.780 (4.981) | -3.766 (9.005) | -3.052 (8.958) | -11.229 (4.218)
  Day 4-Discharge | 6.152 (8.162) | 2.765 (4.557) | -1.697 (4.582) | -1.174 (9.134) | 1.601 (12.279) | -12.798 (3.424)

5. Secondary Outcome: Percent Change From Baseline in Serum Phosphorus
Time Frame: Baseline and 30 minutes, 1, 4, 8, 18, 24, 32, 42, 48, and 56 hours post-dose, and day 4 (discharge).
Population: Participants who were randomized and received any amount of study medication with available data at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pooled Placebo | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide 20 mg | Etelcalcetide 40 mg | Etelcalcetide 60 mg
Number analyzed (Participants) | 20 | 4 | 3 | 4 | 4 | 4
percent change
  30 Minutes: number analyzed (Participants) | 19 | 4 | 3 | 4 | 4 | 4
  30 Minutes | 6.453 (10.400) | 2.080 (4.235) | -0.255 (12.843) | 5.498 (1.546) | 9.024 (10.125) | 5.608 (4.474)
  1 Hour | 10.907 (10.912) | 8.750 (5.519) | 2.219 (15.246) | 12.164 (5.483) | 11.018 (5.492) | 8.621 (4.780)
  4 Hours | 34.009 (16.904) | 34.441 (12.211) | 15.334 (4.080) | 29.231 (15.513) | 30.927 (8.124) | 19.261 (9.807)
  8 Hours | 51.998 (27.762) | 41.575 (33.433) | 9.325 (5.563) | 27.684 (12.520) | 30.640 (24.248) | 32.465 (15.418)
  18 Hours | 69.207 (41.794) | 62.681 (26.476) | 9.206 (2.538) | 30.352 (22.143) | 32.018 (14.688) | 26.240 (19.622)
  24 Hours | 69.676 (45.038) | 55.497 (29.444) | -0.574 (8.659) | 32.376 (28.527) | 24.240 (37.457) | 24.655 (27.651)
  32 Hours | 81.616 (48.245) | 67.662 (43.365) | 12.914 (6.547) | 29.678 (15.174) | 32.705 (28.481) | 43.411 (19.010)
  42 Hours | 82.478 (44.276) | 72.340 (35.380) | 15.357 (8.616) | 35.259 (31.535) | 43.149 (25.219) | 36.299 (31.742)
  48 Hours | 80.245 (48.363) | 66.536 (45.455) | 10.970 (11.808) | 34.452 (31.330) | 43.624 (29.435) | 55.718 (35.112)
  56 Hours: number analyzed (Participants) | 20 | 3 | 3 | 4 | 4 | 4
  56 Hours | 83.741 (51.885) | 98.775 (67.669) | 17.867 (18.308) | 35.569 (21.851) | 43.033 (33.634) | 63.990 (28.031)
  Day 4-Discharge | 83.535 (44.193) | 78.775 (45.141) | 23.022 (12.403) | 54.242 (30.386) | 59.563 (19.668) | 56.708 (29.407)

6. Secondary Outcome: Percent Change From Baseline in Calcium Phosphorus Product
Time Frame: Baseline and 30 minutes, 1, 4, 8, 18, 24, 32, 42, 48, and 56 hours post-dose, and day 4 (discharge).
Population: Participants who were randomized and received any amount of study medication with available data at each time point.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pooled Placebo | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide 20 mg | Etelcalcetide 40 mg | Etelcalcetide 60 mg
Number analyzed (Participants) | 20 | 4 | 3 | 4 | 4 | 4
percent change
  30 Minutes: number analyzed (Participants) | 19 | 4 | 3 | 4 | 4 | 4
  30 Minutes | 6.658 (13.202) | 2.064 (2.420) | -2.929 (14.665) | 2.755 (1.384) | 8.239 (7.640) | 7.789 (10.252)
  1 Hour | 10.828 (14.550) | 8.996 (4.743) | -2.861 (16.546) | 9.236 (4.347) | 6.825 (4.170) | 12.464 (12.914)
  4 Hours | 34.681 (17.635) | 29.766 (10.970) | 6.392 (6.138) | 21.940 (13.151) | 26.340 (10.814) | 17.068 (5.053)
  8 Hours | 53.138 (26.860) | 31.981 (22.948) | -2.240 (9.168) | 17.850 (11.838) | 23.291 (26.675) | 26.854 (17.662)
  18 Hours | 75.585 (43.897) | 57.263 (23.373) | 0.424 (6.565) | 17.405 (17.156) | 24.889 (24.901) | 19.266 (24.212)
  24 Hours | 77.196 (51.499) | 50.020 (23.032) | -9.383 (7.930) | 17.795 (29.202) | 14.095 (38.924) | 18.115 (30.774)
  32 Hours | 87.730 (51.888) | 62.691 (32.631) | 2.355 (8.476) | 16.331 (21.671) | 25.814 (39.166) | 33.902 (27.795)
  42 Hours | 88.570 (48.114) | 62.568 (28.246) | 5.055 (11.224) | 19.449 (29.865) | 30.694 (30.875) | 25.046 (36.401)
  48 Hours | 86.563 (54.601) | 60.665 (40.658) | 0.863 (10.875) | 22.253 (33.958) | 32.771 (35.019) | 39.450 (37.876)
  56 Hours: number analyzed (Participants) | 20 | 3 | 3 | 4 | 4 | 4
  56 Hours | 88.531 (59.100) | 93.793 (59.933) | 5.483 (15.538) | 23.351 (25.107) | 31.825 (42.108) | 44.582 (33.182)
  Day 4-Discharge | 86.989 (50.373) | 73.284 (46.188) | 13.653 (8.448) | 39.885 (28.446) | 46.724 (26.569) | 36.351 (30.774)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Etelcalcetide
Time Frame: Pre-dose and at 0.17, 0.5, 1, 4, 8, 18, 24, 32, and 48 hours after study drug administration and prior to discharge from the clinical research unit (~65 hours).
Population: Participants who were randomized and received any amount of etelcalcetide.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide 20 mg | Etelcalcetide 40 mg | Etelcalcetide 60 mg
Number analyzed (Participants) | 4 | 3 | 4 | 4 | 4
μg/L | 145 (64.8) | 263 (67.2) | 511 (230) | 726 (278) | 1140 (428)

8. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 65 Hours Post-dose for Etelcalcetide
Time Frame: as for outcome 7
Population: Participants who were randomized and received any amount of etelcalcetide with available data.
Measure: Mean (Standard Deviation); unit: hr*μg/L
Arm/Group | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide 20 mg | Etelcalcetide 40 mg | Etelcalcetide 60 mg
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 4
hr*μg/L | 1110 (182) | 2820 (458) | 4920 (1650) | 9560 (3340) | 15700 (5100)

9. Secondary Outcome: Observed Area Under the Concentration-time Curve Extrapolated to Infinity (AUCINFobs) for Etelcalcetide
Time Frame: as for outcome 7
Population: Participants who were randomized and received any amount of etelcalcetide and with available data; The half-life associated with the terminal (log-linear) elimination phase values for the 40 mg dose level were not calculated due to poor log linear regression of the log concentration versus time profile during the terminal phase (r2 values <0.7).
Measure: Mean (Standard Deviation); unit: hr*μg/L
Arm/Group | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide 20 mg | Etelcalcetide 40 mg | Etelcalcetide 60 mg
Number analyzed (Participants) | 3 | 2 | 2 | 0 | 3
hr*μg/L | 3180 (1350) | 5280 (970) | 16800 (4560) |  | 43800 (16900)

10. Secondary Outcome: Percent AUC Extrapolated to Infinity (AUCINF) Resulting From Extrapolation From 65 Hours Onward for Etelcalcetide
Time Frame: as for outcome 7
Population: Participants who were randomized and received any amount of etelcalcetide and with available data.
Measure: Mean (Standard Deviation); unit: percentage of AUCINF
Arm/Group | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide 20 mg | Etelcalcetide 40 mg | Etelcalcetide 60 mg
Number analyzed (Participants) | 3 | 2 | 4 | 3 | 4
percentage of AUCINF | 64.6 (11.4) | 50.9 (9.55) | 71.7 (5.96) | 60.2 (25.8) | 68.0 (8.24)

ADVERSE EVENTS:
Time Frame: For Cohorts 1 to 3, from administration of study drug up until 21 days after study drug administration; for Cohorts 4 and 5 from administration of study drug until 28 days after study drug administration.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Pooled Placebo | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide 20 mg | Etelcalcetide 40 mg | Etelcalcetide 60 mg
Serious Adverse Events (participants affected / at risk) | 1/20 | 0/4 | 0/3 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/20 | 1/4 | 1/3 | 1/4 | 4/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=20) | Etelcalcetide 5 mg (N=4) | Etelcalcetide 10 mg (N=3) | Etelcalcetide 20 mg (N=4) | Etelcalcetide 40 mg (N=4) | Etelcalcetide 60 mg (N=4)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=20) | Etelcalcetide 5 mg (N=4) | Etelcalcetide 10 mg (N=3) | Etelcalcetide 20 mg (N=4) | Etelcalcetide 40 mg (N=4) | Etelcalcetide 60 mg (N=4)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
INJECTION SITE PRURITUS (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
CALCIUM IONISED DECREASED (Investigations) | 0 | 0 | 1 | 0 | 4 | 2
PARAESTHESIA (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.